CLINICAL TRIAL: NCT05026190
Title: Role of Transrectal-ultrasound in Evaluation of Azoospermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed ElSharkawy, resident of urology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: infertility Azoospermia TRUS
Record Dates: First submitted 2021-08-04; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Infertility Due to Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- azoospermic patients (Other)
  Interventions: Diagnostic Test: transrectal ultrasound

INTERVENTIONS:
Diagnostic Test: transrectal ultrasound — we perform trus to identify the cause of azospermia and its type either obstructive or not

SUMMARY:
Azoospermia is a word meaning to ejaculates with no spermatozoa without a definite underlying cause .1% of men has azoospermia, representing nearly 10 to 15% of all infertile men. The azoospermia is a major concern in our community. There is no actual epidemiological studies to estimate the actual numbers in Egypt. Azoospermia has several classifications, pre-testicular, testicular & post-testicular cause .The semen analysis is the main investigation done for these patient .The treatment methods range from hormonal therapy to surgery or ICSI . The imaging modalities has developed greatly in the last 3 decades. That it became in several setting as a bedside test or investigation. The main modalities used in azoospermia are scrotal ultrasound, TRUS and MRI. The first TRUS was introduced 1957.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients with azoospermia as identified by semen analysis.

  * Age from 18 years to more

Exclusion Criteria:

* • History of operative intervention in the lower urinary tract.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2021-10-05 (Estimated); Primary Completion 2022-12-05 (Estimated); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients With obstructive azoospermia | through study completion ,within average one year.
Number of patient with non obstructive azoospermia | through study completion , within average one year.
Number of patient that will respond to endoscopic treatment | 6 month duration
Number of patients that will need sperm extraction | 9 month duration

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aziz N. The importance of semen analysis in the context of azoospermia. Clinics (Sao Paulo). 2013;68 Suppl 1(Suppl 1):35-8. doi: 10.6061/clinics/2013(sup01)05. PMID 23503953
- [Background] Gudeloglu A, Parekattil SJ. Update in the evaluation of the azoospermic male. Clinics (Sao Paulo). 2013;68 Suppl 1(Suppl 1):27-34. doi: 10.6061/clinics/2013(sup01)04. PMID 23503952
- [Background] Cocuzza M, Alvarenga C, Pagani R. The epidemiology and etiology of azoospermia. Clinics (Sao Paulo). 2013;68 Suppl 1(Suppl 1):15-26. doi: 10.6061/clinics/2013(sup01)03. PMID 23503951
- [Background] Sihag P, Tandon A, Pal R, Jain BK, Bhatt S, Kaur S, Sinha A. Sonography in male infertility: a look beyond the obvious. J Ultrasound. 2018 Sep;21(3):265-276. doi: 10.1007/s40477-018-0294-5. Epub 2018 Mar 28. PMID 29594932